CLINICAL TRIAL: NCT04756843
Title: Early Versus Late Orthodontic Treatment of Dental Crowding - a Randomised Controlled Trial
Brief Title: Early Orthodontic Treatment of Dental Crowding
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: City of Vantaa (Other Government)
Responsible Party: Principal Investigator, Heidi Arponen, Principal investigator, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS/3102/2020
Record Dates: First submitted 2021-02-08; First posted 2021-02-16 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Dental Crowding
MeSH Terms: conditions — Crowding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early treatment (Experimental): Treatment started in the early mixed dentition phase
  Interventions: Device: Quad-helix
- Late treatment (Experimental): Treatment started in the late mixed dentition phase
  Interventions: Device: Quad-helix

INTERVENTIONS:
Device: Quad-helix — Fixed orthodontic appliance

SUMMARY:
Aim of the study is to compare treatment duration and effects of orthodontic treatment of dental crowding between treatments started at different stages of mixed dentition phase. The randomized controlled trial study will be conducted in a public health care center.

ELIGIBILITY:
Inclusion Criteria:

* Dental developmental stage of mixed dentition
* Crowding on both dental arches
* Skeletal discrepancy not suspected

Exclusion Criteria:

* National criteria for publicly funded treatment not met by the severity of the malocclusion
* Other malocclusions
* Angle Class III relationship of the molars
* Malocclusion related to a syndrome
* Non-compliance to orthodontic treatment

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Treatment time | Up to 36 months
  Duration of treatment

SECONDARY OUTCOMES:
Treatment burden | Up to 48 months
  Number of orthodontic appliances used
Alignment of dental arches | up to 48 months
  Occlusal end result of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Arponen, DDS, Principal Investigator — University of Helsinki
Locations (1):
- University of Helsinki, Helsinki, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No